CLINICAL TRIAL: NCT05460988
Title: "Re-instrumentation vs Flap Surgery in Residual Pockets: a RCT on Clinical Efficacy"
Brief Title: "Re-instrumentation vs Flap Surgery"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Luigi Barbato, Clinical professor and principal investigator, University of Florence
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18876
Record Dates: First submitted 2022-07-12; First posted 2022-07-15 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Periodontal Pocket; Periodontitis
Keywords: non-surgical periodontal therapy; re-instrumentation
MeSH Terms: conditions — Periodontal Pocket; Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non surgical re-instrumentation (Experimental): The sites showing remaining pockets (PD>4mm), in the sextants allocated to re-instrumentation group, will be treated with subgingival debridement. The subgingival debridement will be performed after the administration of local oral anaesthesia (Articaine 1:100000) using a periodontal tip on ultrasonic instrument (EMS) and Gracey's curettes.
  Interventions: Procedure: Non surgical re-instrumentation
- Flap surgery (Active Comparator): All the sites showing a residual pocket in a sextant allocated to surgery group will receive flap surgery. After the administration of oral local anaesthesia (Articaine 1:100000) an intrasulcular flap will be raised. In order to preserve interdental tissue the flaps will be designed accordingly the principles of papillary preservation flap. Toot root will be carefully debrided using both ultrasonic instruments and Grecey's curettes. Bone recontouring and ostectomy/osteoplasty will be avoided. Single simple sutures will be used to close the flap (Vicryl 5-0).
  Interventions: Procedure: Flap surgery

INTERVENTIONS:
Procedure: Flap surgery — All the sites showing a residual pocket in a sextant allocated to surgery group will receive flap surgery. After the administration of oral local anaesthesia (Articaine 1:100000) an intrasulcular flap will be raised. In order to preserve interdental tissue the flaps will be designed accordingly the principles of papillary preservation flap. Toot root will be carefully debrided using both ultrasonic instruments and Grecey's curettes. Bone recontouring and ostectomy/osteoplasty will be avoided. Single simple sutures will be used to close the flap (Vicryl 5-0).
  Arms: Flap surgery
Procedure: Non surgical re-instrumentation — The sites showing remaining pockets (PD>4mm), in the sextants allocated to re-instrumentation group, will be treated with subgingival debridement. The subgingival debridement will be performed after the administration of local oral anaesthesia (Articaine 1:100000) using a periodontal tip on ultrasonic instrument (EMS) and Gracey's curettes.
  Arms: Non surgical re-instrumentation

SUMMARY:
There are no studies comparing reinstrumentation and flap surgery for the treatment of residual periodontal pockets.

The aim of this RCT is to compare the re-instrumentation vs the flap surgery in terms of PD reduction, CAL gain, gingival recession, need of an additional surgery and pocket closure. Moreover, PROMs will be evaluated

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18aa
* Patients with periodontal disease
* Less than 20 cigarettes/day
* No systemic antibiotic therapy in the last 3 months
* At least one interdental site showing PD≥5mm after the non surgical periodontal initial therapy. Infrabony component of the defect ≤3mm at x-ray
* Full-mouth plaque score and full-mouth bleeding score <15% at baseline (re-evaluation) measured at six sites per tooth
* No previous periodontal surgery at the experimental tooth

Exclusion Criteria:

* Connective tissue diseases
* Diabetes
* Pregnancy or lactating
* Furcation involvement
* Crowned tooth
* Severe tooth mobility (class III)
* Radiographical horizontal bone resorption exceeding the 50% of the root

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
PD change | 3 months after the procedure
  change in periodontal probing depth (in mm)
PD change | 6 months after the procedure
  change in periodontal probing depth (in mm)
PD change | 12 months after the procedure
  change in periodontal probing depth (in mm)

SECONDARY OUTCOMES:
CAL change | 3 months after the procedure
  change in clinical attachment level (in mm)
CAL change | 6 months after the procedure
  change in clinical attachment level (in mm)
CAL change | 12 months after the procedure
  change in clinical attachment level (in mm)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florence, Florence, Florence, Italy

REFERENCES:
- [Derived] Barbato L, Noce D, Di Martino M, Castelluzzo W, Spoleti F, Rupe C, Nieri M, Cairo F. Non-surgical retreatment versus papillary preservation flap surgery for residual pockets: A randomized controlled trial with clinical and patient-reported outcomes. J Clin Periodontol. 2024 Oct;51(10):1277-1288. doi: 10.1111/jcpe.14047. Epub 2024 Jul 16. PMID 39011585